CLINICAL TRIAL: NCT00872326
Title: Phase I/II Study of Regenerative Cell Therapy in Treating Diabetic Patients With Critical Limb Ischemia
Brief Title: Autologous Bone Marrow Derived Mononuclear Cells in Treating Diabetic Patients With Critical Limb Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C/ICPD/2007; FPS C/ICPD/2007
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Peripheral Vascular Diseases; Diabetic Foot
Keywords: Diabetes Complications; Lower limb ischemia; Adult stem cells
MeSH Terms: conditions — Peripheral Vascular Diseases; Diabetic Foot; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Bone Marrow Mononuclear Cells (Experimental): Consecutive inclusion among diabetic patients with critical limb ischemia. Intraarterial infusion of autologous bone marrow mononuclear cells
  Interventions: Procedure: Autologous Bone Marrow Mononuclear Cells

INTERVENTIONS:
Procedure: Autologous Bone Marrow Mononuclear Cells — Infusion > 80 millions mononuclear cells. Intraarterial administration at popliteal artery level. Infusion during 3 minutes with antegrade blockage of arterial flow.

SUMMARY:
The aim of this study is to assess the efficacy and safety of autologous transplantation of bone-marrow cells for therapeutic angiogenesis and vasculogenesis in diabetic patients with non-revascularizable critical limb ischemia.

DETAILED DESCRIPTION:
Phase I/II, prospective, single-center study, with consecutive inclusion of 20 diabetic patients with critical limb ischemia due to bellow-the-knee extensive arterial disease.

After the inclusion, patients are submitted to a bone-marrow aspiration (30 ml) under sedation. Autologous bone-marrow mononuclear cells (minimum 80 millions mononuclear cells) are infused intraarterially at popliteal artery by blocking antegrade perfusion during 3 minutes.

Clinical and angiographic follow-up will be performed at 3 months after the infusion to assess the efficacy of autologous mononuclear cells transplantation in terms of:

* Changes in below-the-knee angiography from baseline to 3 months follow-up.
* Changes in Ankle-Brachial pressure Index, transcutaneous oxygen pressure, and size of main ischemic ulcer will be also assessed at target limb.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients under treatment (type I or II)
* Critical limb ischemia (rest pain and/or non-healing ischemic ulcers lasting more than 4 weeks, and/or Ankle-Brachial Index < 0,8)
* Not suitable to be revascularized (surgical and interventional consensus)

Exclusion Criteria:

* Neoplastic disease and/or hematologic disease during the last 2 years
* Diabetic retinopathy
* Ischemic ulcer greater than 10 cm2
* Major amputation at target limb
* Life expectancy > 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Angiographic evaluation of angiogenesis and vasculogenesis at target limb | 3 months

SECONDARY OUTCOMES:
Ankle-Brachial pressure index | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio de la Cuesta, MD, Principal Investigator — Critical Limb Ischemia Unit. Hospital Universitario Virgen Macarena and Hospital San Lazaro; Manuel Constantino, PhD, Principal Investigator — Chief of Hematology. Hospital Universitario Virgen Macarena; Rafael J Ruiz-Salmeron, PhD, Principal Investigator — Chief of Endovascular Unit. Hospital Universitario Virgen Macarena
Locations (1):
- University Hospital Virgen Macarena, Seville, Seville, Spain

REFERENCES:
- [Derived] Ruiz-Salmeron R, de la Cuesta-Diaz A, Constantino-Bermejo M, Perez-Camacho I, Marcos-Sanchez F, Hmadcha A, Soria B. Angiographic demonstration of neoangiogenesis after intra-arterial infusion of autologous bone marrow mononuclear cells in diabetic patients with critical limb ischemia. Cell Transplant. 2011;20(10):1629-39. doi: 10.3727/096368910X0177. PMID 22289660